CLINICAL TRIAL: NCT03960749
Title: The Importance of Needle Size, Needle Design and Stylet Reinsertion to Prevent Post-lumbar Puncture Headache, a Randomized Controlled Trial
Brief Title: Headache After Diagnostic Lumbar Puncture
Acronym: HELPUmeå
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonatan Salzer (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Jonatan Salzer, Principal Investigator, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HELP Umeå
Record Dates: First submitted 2019-05-02; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Post-Lumbar Puncture Headache
Keywords: Lumbar puncture; Headache
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache | interventions — Needles

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group. Randomization between three different lumbar puncture needles and between stylet reinsertion of not before needle withdrawal.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are not informed about the allocated needle. The follow-up telephone calls (outcome assessment) are made by an assistant nurse who is unaware of randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sprotte 25G needle, stylet reinserted (Experimental)
  Interventions: Device: Sprotte 25G needle, stylet reinserted
- Sprotte 25G needle, stylet not reinserted (Experimental)
  Interventions: Device: Sprotte 25G needle, stylet not reinserted
- Sprotte 22G needle, stylet reinserted (Experimental)
  Interventions: Device: Sprotte 22G needle, stylet reinserted
- Sprotte 22G needle, stylet not reinserted (Experimental)
  Interventions: Device: Sprotte 22G needle, stylet not reinserted
- Spinocan 25G needle, stylet reinserted (Experimental)
  Interventions: Device: Spinocan 25G needle, stylet reinserted
- Spinocan 25G needle, stylet not reinserted (Experimental)
  Interventions: Device: Spinocan 25G needle, stylet not reinserted

INTERVENTIONS:
Device: Sprotte 25G needle, stylet reinserted — Lumbar puncture with small bore atraumatic needle, stylet reinserted before needle withdrawal
  Arms: Sprotte 25G needle, stylet reinserted
Device: Sprotte 25G needle, stylet not reinserted — Lumbar puncture with small bore atraumatic needle, stylet not reinserted before needle withdrawal
  Arms: Sprotte 25G needle, stylet not reinserted
Device: Sprotte 22G needle, stylet reinserted — Lumbar puncture with larger bore atraumatic needle, stylet reinserted before needle withdrawal
  Arms: Sprotte 22G needle, stylet reinserted
Device: Sprotte 22G needle, stylet not reinserted — Lumbar puncture with larger bore atraumatic needle, stylet not reinserted before needle withdrawal
  Arms: Sprotte 22G needle, stylet not reinserted
Device: Spinocan 25G needle, stylet reinserted — Lumbar puncture with small bore cutting needle, stylet reinserted before needle withdrawal
  Arms: Spinocan 25G needle, stylet reinserted
Device: Spinocan 25G needle, stylet not reinserted — Lumbar puncture with small bore cutting needle, stylet not reinserted before needle withdrawal
  Arms: Spinocan 25G needle, stylet not reinserted

SUMMARY:
The objectives of this study are to investigate the effects of needle design, needle size and stylet reinsertion on the risk for headache after diagnostic LP (lumbar puncture, Post-LP headache). The following needles are used in the study:

1. Sprotte 25 Gauge (G) (0.5 mm) atraumatic needle with introducer
2. Sprotte 22 G (0.7 mm) atraumatic needle with introducer
3. Spinocan 25 G (0.5 mm) cutting needle

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing diagnostic LP during their neurological work-up at Umeå University Hospital, Sweden, from 28 May 2013 until the study is fully recruited and;
* Willing to participate and
* Providing informed consent

Exclusion Criteria:

-Subjects unable to participate in the study follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Odds ratio for post-lumbar puncture headache (any) | Up to 14 days after LP
  Any post-lumbar puncture headache (as defined in the international classification of headache disorders 3 (ICHD-3).

SECONDARY OUTCOMES:
Odds ratio for post-lumbar puncture headache (severe) | Up to 14 days after LP
  Severe (preventing daily activities) post-lumbar puncture headache (as defined in the international classification of headache disorders 3 (ICHD-3).
Headache duration (days) | Until cessation, up to 14 days after LP
Proportion using analgesia | During post-lumbar puncture headache, up to 14 days after LP
Proportion on sick leave | During post-lumbar puncture headache, up to 14 days after LP
Proportion with back pain | Up to 14 days after LP
Proportion with radiating leg pain | Up to 14 days after LP
Multiplicative interactions between age (years), sex, BMI and needle visavi the outcome "any post-LP headache" in a multivariable logistic regression model | Up to 14 days after LP
  Interactions between important predictors of headache and needle allocation, assessed in multivariable logistic regression models with interaction terms which are the products of the two potentially interacting variables. Age and BMI will be treated as continuous variables, sex and needle allocation as categorical variables.

OTHER OUTCOMES:
Procedure duration (minutes) | During the lumbar puncture
  Procedure duration from start of procedure (defined as when the operator starts palpating the iliac crest) until procedure cessation (defined as when the needle is withdrawn from the participant).
Proportion undergoing needle switch | During the lumbar puncture
  Technical difficulties may differ between needles and thus the proportion undergoing needle switch due to these difficulties may differ.
Opening pressure (cm H2O) | During the lumbar puncture
  Opening pressure measured immediately after cerebrospinal fluid (CSF) contact using a thin tube attached to a paper ruler, using the skin entry hole as reference point. This is only performed in the recumbent position.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans RW, Armon C, Frohman EM, Goodin DS. Assessment: prevention of post-lumbar puncture headaches: report of the therapeutics and technology assessment subcommittee of the american academy of neurology. Neurology. 2000 Oct 10;55(7):909-14. doi: 10.1212/wnl.55.7.909. No abstract available. PMID 11061243
- [Background] Hyllienmark L, Zachau AC. [Diagnostic lumbal puncture]. Lakartidningen. 2008 Oct 8-14;105(41):2844-9. No abstract available. Swedish. PMID 19009898
- [Background] Armon C, Evans RW; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Addendum to assessment: Prevention of post-lumbar puncture headaches [RETIRED]: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2005 Aug 23;65(4):510-2. doi: 10.1212/01.wnl.0000173034.96211.1b. PMID 16116106
- [Background] Strupp M, Brandt T. Should one reinsert the stylet during lumbar puncture? N Engl J Med. 1997 Apr 17;336(16):1190. doi: 10.1056/NEJM199704173361616. No abstract available. PMID 9102578
- [Background] Hammond ER, Wang Z, Bhulani N, McArthur JC, Levy M. Needle type and the risk of post-lumbar puncture headache in the outpatient neurology clinic. J Neurol Sci. 2011 Jul 15;306(1-2):24-8. doi: 10.1016/j.jns.2011.04.004. Epub 2011 May 5. PMID 21549395
- [Background] Strupp M, Schueler O, Straube A, Von Stuckrad-Barre S, Brandt T. "Atraumatic" Sprotte needle reduces the incidence of post-lumbar puncture headaches. Neurology. 2001 Dec 26;57(12):2310-2. doi: 10.1212/wnl.57.12.2310. PMID 11756618

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03960749/Prot_SAP_000.pdf